CLINICAL TRIAL: NCT06208787
Title: Combining Novel Bio-Neurofeedback Techniques With Mindfulness-Based Interventions to Reduce Symptoms of Mental Distress
Brief Title: Neurofeedback-Assisted Mindfulness Techniques to Reduce Symptoms of Mental Distress
Acronym: ComBiNe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Alaerts, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S68049
Record Dates: First submitted 2023-12-21; First posted 2024-01-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Stress
Keywords: neurofeedback; mindfulness; stress; cross-frequency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Individuals assigned to this group will receive the experimental neurofeedback training
  Interventions: Behavioral: Neurofeedback training
- Control group (Sham Comparator): Individuals assigned to this group will receive the sham neurofeedback training
  Interventions: Behavioral: Sham Training

INTERVENTIONS:
Behavioral: Neurofeedback training — Neurofeedback training involving auditory feedback upon measurement of non-harmonic alpha-theta ratios during focused attention meditation
  Arms: Experimental group
Behavioral: Sham Training — Sham neurofeedback involving auditory feedback at random timepoints during focused attention meditation such that no learning can take place
  Arms: Control group

SUMMARY:
Neurofeedback training, based on operant conditioning techniques, involves the measurement and conscious regulation of specific neural parameters through participant-specific feedback. This technique has gained recognition for its role in efficiently altering brain activity. Among its various applications, neurofeedback training is noted for its ability to facilitate meditative practice and enhance stress regulation abilities. However, most neurofeedback studies focus on modulating isolated brainwaves and overlook how brainwaves interact across frequencies. To address this gap, the present study will evaluate an intervention that combines meditation techniques with a novel cross-frequency neurofeedback training to enhance the outcomes of meditative practice for stress regulation.

Previous research has established that brain rhythms exhibit interactive patterns, forming harmonic and non-harmonic relationships to respectively facilitate and preclude cross-frequency coupling. Harmonic relationships are essential for the synchronization of oscillations, a process necessary for coordinating complex neural and physiological activities. In contrast, non-harmonic relationships result in a highly desynchronized state characterized by reduced neural and physiological coordination, typically observed during cognitive restful periods. In this regard, prior studies have demonstrated a link between an increased occurrence of non-harmonic alpha-theta ratios and mindfulness meditation.

Recent research has shown the possibility of upregulating the incidence of non-harmonic alpha-theta ratios during mindfulness meditation in a single-session neurofeedback training context. However, the impact of long-term training on stress regulation abilities remains unclear. The current study addresses this gap by conducting a 10-session neurofeedback training focused on upregulating the incidence of non-harmonic alpha-theta ratios during focused attention meditation. The primary aim of this study is to determine the effectiveness of this training in assisting mindfulness practice and improving stress regulation as assessed by a range of neurophysiological, psychological, and biological outcomes.

DETAILED DESCRIPTION:
The present study is a single-blind, randomized-controlled clinical trial involving 80 healthy, meditation-naïve adults. All participants will be randomly assigned to either take part in experimental neurofeedback training or control (sham) neurofeedback training. Each training consists of 10 training sessions, with a frequency of 2 sessions per week (i.e., 5 weeks total training duration).

During each neurofeedback training session, participants will sit in front of a computer screen in a dimly lit room. Each training session will start and finish with a self-report mood assessment (POMS) and a 2-minute neural resting-state recording. In-between, participants will take part in 10 consecutive 2-minute neurofeedback trials. During these trials, participants are instructed to close their eyes and focus their attention on a specific point of their body (i.e., an anchor point). Simultaneously, neural recordings will be made, and reinforcing auditory cues will be presented upon the measurement of non-harmonic ratios between alpha and theta rhythms at the Pz channel. Participants are informed that the feedback sounds serve as positive feedback for their ability to engage in a neurophysiological state associated with meditative practice for stress regulation, and that this sound will assist their body in self-regulating to sustain this desired state. The sham training will be indistinguishable from the experimental biofeedback training for the participants involved. However, during the sham training, auditory cues will be unrelated to the participant's underlying brain activity, presented at random timepoints and therefore, no specific training can occur. After every two training trials, participants will be asked to indicate their levels of focus, sleepiness, and relaxation.

The investigators will measure psychological, neurophysiological, and biological mental health outcomes before the start of the training (T0), following the end of the training (T1), and again at the 5-week follow-up (T2).

During these three assessment points, participants will complete self-report questionnaires on emotional distress (DASS), mindfulness skills (CHIME), perceived stress (PSS), repetitive negative thinking (PTQ), and sleep quality (PSQI). Next, neurophysiological measurements will be made during a 5-minute eyes-closed resting state recording, during a 10-minute eyes-closed focused attention meditation, and during eyes-closed stress induction (3 min) and recovery (17 out of 57 min). Stress will be induced by utilizing the cold pressor task procedure which involves the participant submerging their hand into cold water (0-2°C) for a duration of three minutes while being perceived to be recorded by a video camera. Cortisol samples will be obtained right before the stress induction (T0), during the expected cortisol peak (T0 + 20 minutes) and after a recovery period (T0 + 60 minutes).

In addition, the day following each assessment session, participants will be asked to apply mobile health patches for ambulant recording of their cardiac activity for a duration of 24 hours. At the same time, stress reactivity in daily life will be assessed using the experience sampling method. To this end, participants will be prompted on their smartphones at semi-random moments during the daytime to indicate how they are feeling for 4 consecutive days (10 prompts per day). Finally, in the morning of each assessment day, participants will collect salivary samples for the assessment of cortisol and oxytocin levels.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent;
* Dutch or English speaking;
* Experience mild to severe stress symptoms (as measured by a score between 15 and 33 on the Stress Subscale of the DASS-21).

Exclusion Criteria:

* History of psychotropic medication usage in the past six months;
* Substantial experience with meditative practices (including but not limited to mindfulness, yoga, tai chi, or other similar practices) by meeting any of the following criteria:

  1. Participant has participated in a multi-day meditation retreat or program during the past year;
  2. Participant engages in meditative practices on a weekly basis or more frequently, for at least six consecutive weeks, within six month prior to the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
occurrence of non-harmonic alpha-theta ratios at rest | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  EEG recording
occurrence of non-harmonic alpha-theta ratios during meditation | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  EEG recording
occurrence of non-harmonic alpha-theta ratios during stress induction | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  EEG recording
occurrence of non-harmonic alpha-theta ratios during stress recovery | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  EEG recording
self-reported levels of emotional distress | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  DASS questionnaire

SECONDARY OUTCOMES:
self-reported levels of mindfulness skills | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  CHIME questionnaire
self-reported levels of perceived stress | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  PSS questionnaire
self-reported levels of repetitive negative thinking | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  PTQ questionnaire
self-reported levels of sleep quality | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  PSQI questionnaire

OTHER OUTCOMES:
salivary oxytocin levels | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  saliva sample (exploratory)
salivary cortisol levels | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  saliva sample (exploratory)
mood in daily life | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  experience sampling method (exploratory)
cardiac activity in the lab | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  ECG recording (exploratory)
cardiac activity in daily life | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  ECG recording (exploratory)
respiratory activity in the lab | pre-intervention (week 0), post-intervention (week 6), follow-up (week 11)
  respiration recording (exploratory)
mood state during training sessions | during each training session (i.e., twice during week 1, 2, 3, 4, and 5)
  POMS questionnaire + single items (fatigue, focus, sleepiness) (exploratory)

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Alaerts, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No